CLINICAL TRIAL: NCT05019196
Title: Neuroimaging Study on the Recombination of Brain Motor and Language Function Induced by Glioma
Brief Title: fMRI Study of Functional Reorganization in Glioma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018SF-113
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-08

CONDITIONS: Glioma
Keywords: low-grade glioma; fMRI; function reorganization
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fMRI，functional reorganization, functional connectivity, functional rating scale: low-grade glioma patients healthy controls
  Interventions: Device: GE 3.0T MRI

INTERVENTIONS:
Device: GE 3.0T MRI — using GE 3.0T MRI to obtain anatomical and functional MR images and DTI images

SUMMARY:
Glioma is an invasive growth, easy to relapse, poor prognosis, great harm to human and society. Studies have shown that gliomas can cause the dynamic reorganization of brain functional areas, affecting the accuracy of surgical resection and the evaluation of long-term efficacy. While, it is difficult to monitor the functional reorganization of glioma in existing studies. The development trend can not effectively predict the outcome of tumor anaplasia and the compensation of brain function, which restricts the accurate tumor resection. In the early stage of this study, functional connectivity analysis was carried out of gliomas in the motor region and showed that the damage of motor functional connectivity on the opposite side of the lesion occurred earlier than that on the same side, suggesting that there may be some rules of how the disease caused functional reorganization. After stroke, the language and motor function will undergo plasticity, causing the functional areas to slowly repair the damaged function. Contrast to stroke, low-grade glioma grows slower, which gives brain more time to adapt to the damage caused by tumor growth, it may cause more functional reorganization. Professor Hugues Duffau's research showed that it is brain plasticity that can effectively explain patients with low-grade gliomas, even in language and motor areas, did not appear obvious dysfunction. Our previous research found there were significant differences in motor functional connectivity between the two hemispheres of the patients between the plasma tumor group and healthy controls. In addition, in the tumor group, the damage of motor connection on the contralateral side of the lesion occurred before on the ipsilateral side. These results suggest that brain function has been remodeled in patients with brain tumors who have not yet exhibited motor impairment. We presume there may be a certain pattern of brain function reorganization caused by low-grade glioma. This study take patients with brain glioma as the research object and adopt a multi-time point experimental design, combining with cortical electrical stimulation and multimodal magnetic resonance imaging data before and after operation, intending to observe the dynamic changes of language and motor function networks.

DETAILED DESCRIPTION:
Glioblastoma is the most common malignant tumor of the central nervous system in adults. It is highly invasive, grows rapidly and has a poor prognosis. Brain tumors, whether benign or malignant in nature, take up space in the skull and will follow the tumor. The malignant degree of growth, so that the intracranial pressure increases, thus compression or destruction of brain tissue, leading to central nervous damage, it endangers the life of the patient.

At present, neurosurgery is still the main treatment for craniocerebral tumors. Surgical resection course degree is a determinant of patient survival. Due to individual differences and pathological changes, the effect of causing the variation of the anatomical position of brain functional areas and the generation of intraoperative brain tissue displacement all make it difficult to determine correct functional areas, which is the main reason that affects the accuracy and postoperative effect of surgery.

However, routine MRI scans have difficulty in identifying changes in adjacent functional areas caused by tumors, and is also difficult to define the boundaries of invasive neoplasms. The application of functional magnetic resonance imaging and diffusion tensor imaging enables neurosurgeons not only to be accurate positioning the functional areas, but knowing the functional areas caused by the tumor before neurosurgery, so as to maximize removing the tumor and better protecting important functional areas.

After stroke, the language and motor function will undergo plasticity, causing the language and motor areas to slowly repair the damaged brain function. Contrast to stroke, low-grade glioma grows slower, which gives brain more time to adapt to the damage caused by tumor growth, it may cause more functional reorganization. Professor Hugues Duffau's research, published in the journal Brain, also shows that it is brain plasticity that can effectively explain patients with low-grade gliomas, even in language and motor areas, did not appear obvious dysfunction. Therefore, exploring the brain functional plasticity of low-grade glioma not only facilitates the maximum resection of the tumor, but also help for prediction of postoperative of rehabilitation.

Therefore, taking the patients with brain glioma as the object in this project, combining with intraoperative cortical electrical stimulation and multiple modal magnetic resonance imaging, a multi-time longitudinal study was designed to explore the imaging features of changes in motor and language plasticity in low-grade gliomas.

All images were obtained using a GE3.0T magnetic resonance scanner. 3D-T1FSPGR（ fast spoiled gradient echo）was scanned for anatomical images, T2-weighted single-shot gradient-echo-planae-imaging sequence for functional images. Tak-based fMRI used block design mode (e.g. ABAB mode) with 30s resting state (A) and 30s hand movement task (B) alternating, the whole task process has a total of 6 resting states, 5 tasks state composition. All patients and healthy controls were instructed to repeatedly play each visual stimulus with open and close hand. All the subjects were trained on a specific exercise task before the scans, to ensure that the task is fully understood and that you are able to cooperate carefully to complete the scan. Language tasks use the block design paradigm. The equation is control-task-control last for 5min30s with 30s interval.

In this study, the subjects looked at the "+" symbol on the screen and lay quietly on the exam bed performing three language tasks. All the patients were trained to better cooperate with the subjects. To avoid head movement displacement during scanning, patients are required to speak as softly as possible that is whisper. Furthermore，derect electric stimulus was conducted in every patient. If the distance between functional areas and the positive target of electrical stimulation was less than 1cm, the results of fMRI and electrical considered were considered to be consistent. As for functional rating scale, the standard chinese version of the Quality of Life Inventory EORTC QLQ-C30 (3.0) was used to assess the preoperative quality of life of patients with brain tumors; KPS( Karnofsky Performance Status Scale）was used to evaluate physiological function; Mini-Mental State Examination (MMSE) was used for clinical screening of cognitive impairment, evaluate the patients' interpretation, spatial orientation, memory and computation, linguistic naming and reading ability.

Correlation analysis was conducted between the fMRI data processing results and functional scale score, to build the brain structure - function correlation models and explore different stages of low-grade glioma recombination mode of functional areas.

ELIGIBILITY:
Inclusion Criteria:

* All cases underwent no treatment or surgery before examination;
* Can cooperate to complete routine MRI, fMRI, DTI, and rfMRI were required and the image quality was graded the value of analysis;
* All cases were confirmed by craniotomy and pathology;
* Right-handed;
* Mass lesion located in the left dominant hemisphere
* single lesion;
* No chronic diseases such as hypertension and diabetes

Exclusion Criteria:

* History of neurological diseases;
* Previous history of brain trauma accompanied by consciousness disorder;
* Before scanning 6, a history of long-term use of psychoactive substances such as alcohol and drug within one month;
* Obviously mentally handicapped;
* magnetic resonance (NMR) check for contraindications;
* Family history of neuropsychiatric disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fifty patients with right-handed low-grade glioma who met the inclusion and exclusion criteria were included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of functional connections between cerebral hemispheric regions | 2021.12.1
  This study selected the functional activation regions of the patients' own motor or language tasks were used as seed points for the functional connections of complex brain networks analysis. Each region of interest is defined as a sphere with a radius of 6mm for functional connection analysis. Among them, Pearson's correlation coefficient was used as a pairing calculation between brain regions in each patient. Apply the Fisher's r turnZ method is used to improve the normality of the correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Chen Niu, PhD, Study Director — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marusyk A, Almendro V, Polyak K. Intra-tumour heterogeneity: a looking glass for cancer? Nat Rev Cancer. 2012 Apr 19;12(5):323-34. doi: 10.1038/nrc3261. PMID 22513401
- [Result] Stupp R, Brada M, van den Bent MJ, Tonn JC, Pentheroudakis G; ESMO Guidelines Working Group. High-grade glioma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii93-101. doi: 10.1093/annonc/mdu050. Epub 2014 Apr 29. No abstract available. PMID 24782454
- [Result] Rosler J, Niraula B, Strack V, Zdunczyk A, Schilt S, Savolainen P, Lioumis P, Makela J, Vajkoczy P, Frey D, Picht T. Language mapping in healthy volunteers and brain tumor patients with a novel navigated TMS system: evidence of tumor-induced plasticity. Clin Neurophysiol. 2014 Mar;125(3):526-36. doi: 10.1016/j.clinph.2013.08.015. Epub 2013 Sep 16. PMID 24051073
- [Result] Southwell DG, Hervey-Jumper SL, Perry DW, Berger MS. Intraoperative mapping during repeat awake craniotomy reveals the functional plasticity of adult cortex. J Neurosurg. 2016 May;124(5):1460-9. doi: 10.3171/2015.5.JNS142833. Epub 2015 Nov 6. PMID 26544767
- [Result] Duffau H. The huge plastic potential of adult brain and the role of connectomics: new insights provided by serial mappings in glioma surgery. Cortex. 2014 Sep;58:325-37. doi: 10.1016/j.cortex.2013.08.005. Epub 2013 Aug 19. PMID 24050218
- [Result] Saito T, Muragaki Y, Miura I, Tamura M, Maruyama T, Nitta M, Kurisu K, Iseki H, Okada Y. Functional plasticity of language confirmed with intraoperative electrical stimulations and updated neuronavigation: case report of low-grade glioma of the left inferior frontal gyrus. Neurol Med Chir (Tokyo). 2014;54(7):587-92. doi: 10.2176/nmc.cr.2013-0248. Epub 2014 Feb 28. PMID 24584281
- [Result] Duffau H. Lessons from brain mapping in surgery for low-grade glioma: insights into associations between tumour and brain plasticity. Lancet Neurol. 2005 Aug;4(8):476-86. doi: 10.1016/S1474-4422(05)70140-X. PMID 16033690
- [Result] Duffau H. Diffuse low-grade gliomas and neuroplasticity. Diagn Interv Imaging. 2014 Oct;95(10):945-55. doi: 10.1016/j.diii.2014.08.001. Epub 2014 Sep 16. PMID 25218490
- [Result] Briganti C, Sestieri C, Mattei PA, Esposito R, Galzio RJ, Tartaro A, Romani GL, Caulo M. Reorganization of functional connectivity of the language network in patients with brain gliomas. AJNR Am J Neuroradiol. 2012 Nov;33(10):1983-90. doi: 10.3174/ajnr.A3064. Epub 2012 May 3. PMID 22555573
- [Result] Otten ML, Mikell CB, Youngerman BE, Liston C, Sisti MB, Bruce JN, Small SA, McKhann GM 2nd. Motor deficits correlate with resting state motor network connectivity in patients with brain tumours. Brain. 2012 Apr;135(Pt 4):1017-26. doi: 10.1093/brain/aws041. Epub 2012 Mar 8. PMID 22408270
- [Result] Desmurget M, Bonnetblanc F, Duffau H. Contrasting acute and slow-growing lesions: a new door to brain plasticity. Brain. 2007 Apr;130(Pt 4):898-914. doi: 10.1093/brain/awl300. Epub 2006 Nov 21. PMID 17121742
- [Result] Abd-El-Barr MM, Saleh E, Huang RY, Golby AJ. Effect of disease and recovery on functional anatomy in brain tumor patients: insights from functional MRI and diffusion tensor imaging. Imaging Med. 2013 Aug 1;5(4):333-346. doi: 10.2217/iim.13.40. PMID 24660024
- [Result] Tuntiyatorn L, Wuttiplakorn L, Laohawiriyakamol K. Plasticity of the motor cortex in patients with brain tumors and arteriovenous malformations: a functional MR study. J Med Assoc Thai. 2011 Sep;94(9):1134-40. PMID 21970205
- [Result] Kosla K, Pfajfer L, Bryszewski B, Jaskolski D, Stefanczyk L, Majos A. Functional rearrangement of language areas in patients with tumors of the central nervous system using functional magnetic resonance imaging. Pol J Radiol. 2012 Jul;77(3):39-45. doi: 10.12659/pjr.883373. PMID 23049580
- [Result] Bryszewski B, Pfajfer L, Antosik-Biernacka A, Tybor K, Smigielski J, Zawirski M, Majos A. Functional rearrangement of the primary and secondary motor cortex in patients with primary tumors of the central nervous system located in the region of the central sulcus depending on the histopathological type and the size of tumor: Examination by means of functional magnetic resonance imaging. Pol J Radiol. 2012 Jan;77(1):12-20. doi: 10.12659/pjr.882576. PMID 22802861
- [Result] Niu C, Zhang M, Min Z, Rana N, Zhang Q, Liu X, Li M, Lin P. Motor network plasticity and low-frequency oscillations abnormalities in patients with brain gliomas: a functional MRI study. PLoS One. 2014 May 7;9(5):e96850. doi: 10.1371/journal.pone.0096850. eCollection 2014. PMID 24806463
- [Result] Small SL, Buccino G, Solodkin A. Brain repair after stroke--a novel neurological model. Nat Rev Neurol. 2013 Dec;9(12):698-707. doi: 10.1038/nrneurol.2013.222. Epub 2013 Nov 12. PMID 24217509
- [Result] Duffau H. Stimulation mapping of white matter tracts to study brain functional connectivity. Nat Rev Neurol. 2015 May;11(5):255-65. doi: 10.1038/nrneurol.2015.51. Epub 2015 Apr 7. PMID 25848923